CLINICAL TRIAL: NCT06769984
Title: A Multicentre, Randomized, Double-blinded, Placebo-controlled Phase I/II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of SCTT11 in Healthy Participants and Participants with Moderate-to-severe Thyroid Eye Disease
Brief Title: A Study of SCTT11 in Healthy Participants and Participants with Thyroid Eye Disease.
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCTT11-X201
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-12

CONDITIONS: TED

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SCTT11 dose 1, dose 2, dose 3, dose 4 (Experimental)
  Interventions: Drug: SCTT11
- Placebo dose 1, dose 2, dose 3, dose 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SCTT11 — SCTT11 dose 1, dose 2, dose 3, dose 4
  Arms: SCTT11 dose 1, dose 2, dose 3, dose 4
Drug: Placebo — Placebo dose 1, dose 2, dose 3, dose 4
  Arms: Placebo dose 1, dose 2, dose 3, dose 4

SUMMARY:
Multicentre, Randomized, Double-blinded, Phase I/II Clinical Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of SCTT11 in Healthy Participants and Participants with Thyroid Eye Disease

ELIGIBILITY:
Inclusion Criteria for Healthy Participants:

1. Healthy male or female participants aged between18 and 45 inclusive
2. All participants must agree to not fall pregnant and voluntarily use highly effective double method contraception during the study for at least 180 days after the last dose; female participants must have a negative pregnancy test prior to dosing and must not be breastfeeding

Exclusion Criteriafor Healthy Participants:

1.With any other disease or medical condition of clinical significance (e.g., past medical history of chronic hepatic, renal, cardiovascular, neurological/psychiatric, gastrointestinal, respiratory, urological, endocrinological, or other systemic diseases, etc.) as assessed by the investigator.

Inclusion Criteria for TED Participants:

1. Male or female participants aged between 18 and 70 inclusive
2. Participants with moderate-to-severe (has an appreciable impact on daily life and requires intervention, but is not sight-threatening) TED
3. Normal thyroid function, or only mild hyperthyroidism or hypothyroidism (defined as screening free triiodothyronine [FT3] and free thyroxine [FT4] levels < 50% above or below the normal limits).

Exclusion Criteria for TED Participants:

1. Decreased best corrected visual acuity of the study eye due to optic neuropathy within 6 months prior to the first dose
2. Corneal abnormalities in study eye with no relief from treatment, as evaluated by the investigator
3. A reduction of ≥2 points in the CAS value or a reduction of ≥2 mm in proptosis in the study eye from the screening assessment period to study baseline period
4. Presence of other ocular conditions that, in the judgement of the investigator, may affect the evaluation of the study results
5. Presence of poorly controlled diabetes mellitus
6. The current presence of other uncontrolled clinical diseases or conditions
7. Abnormalities in any of the following laboratory examinations during the screening phase
8. Poorly controlled hypertension
9. With past medical histories of major surgery and/or trauma within 1 month prior to the first dose
10. With past medical histories of severe allergies, histories of severe drug allergies, known or suspected allergy to any component of this investigational product
11. Vaccination with live or live attenuated vaccine within 1 month prior to the first dose or expected during the study
12. Participation in a clinical study of any drug or device within 3 months prior to the first dose and have used the investigational product or have been treated with the device
13. Pregnant, lactating females; or participants of childbearing potential who are unwilling to use effective contraception during the study and within 180 days after the last dose
14. Other conditions evaluated by the investigator to be unsuitable for enrolment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-19 (Estimated); Primary Completion 2026-06-24 (Estimated); Study Completion 2028-09-19 (Estimated)

PRIMARY OUTCOMES:
The occurrences of treatment-emergent adverse events (TEAE), treatment-related TEAE (TRAE), serious adverse events (SAE), and adverse events of special interest (AESI) | Day 0 up to 85 days for healthy participants
Proptosis Responder Rate in the study eye | Day 0 up to 169 days
  Proptosis Responder Rate in the study eye (i.e., reduction of proptosis of ≥ 2 mm from baseline without a corresponding increase of ≥ 2 mm in the fellow eye] as measured by exophthalmometer)

SECONDARY OUTCOMES:
Change from baseline in proptosis in the study eye as measured by exophthalmometer | Day 0 up to 169days
Change from baseline in Clinical Activity Score (CAS) | Day 0 up to 169days
Diplopia Responder Rate | Day 0 up to 169days
  Diplopia Responder Rate (i.e., reduction in Gorman Subjective Diplopia Score of ≥1 from baseline for participants with baseline Gorman Subjective Diplopia Score >0)
Proportion of participants with a CAS of zero or one in the study eye | Day 0 up to 169days
SCTT11 concentrations in the blood over time | Day 0 up to 169days
Incidence of anti-drug antibody (ADA) development in SCTT11-treated participants over time | Day 0 up to 169days